CLINICAL TRIAL: NCT01206322
Title: Enhancement of Cerebral Vasoreactivity and Cognition by Intranasal Insulin in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston University (Other); Joslin Diabetes Center (Other); Peking University (Other); University of Washington (Other); University of Arkansas (Other); VA Boston Healthcare System (U.S. Federal Agency); University of Massachusetts, Worcester (Other); Wake Forest University (Other)
Responsible Party: Principal Investigator, Vera Novak, MD PhD, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1R21-DK088446301
Record Dates: First submitted 2010-08-20; First posted 2010-09-21 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes, blood flow, brain perfusion, cognitive function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin vs. placebo (Experimental): Comparisons of acute effects of intranasal insulin or placebo (saline) on cerebral blood flow and cognition in healthy controls and type 2 diabetes.
  Interventions: Drug: Intranasal insulin; Drug: Placebo
- Healthy vs. Diabetic (Other): Comparisons of acute effects of intranasal insulin or placebo (saline) on cerebral blood flow and cognition in healthy controls and type 2 diabetes.
  Interventions: Drug: Intranasal insulin; Drug: Placebo

INTERVENTIONS:
Drug: Intranasal insulin — The acute effects of a single 40-IU dose of intranasal insulin
  Other Names: Novolin R
Drug: Placebo — The acute effects of intranasal sterile saline.

SUMMARY:
Our goal is to determine the acute effects of intranasal insulin on regional perfusion and cognition of older adults. We propose a pilot study to examine the effect of a single dose of intranasal insulin on regional vasoreactivity and cognitive functions in 30 subjects with T2DM and 30 healthy controls >50 years old using a double blinded, placebo-controlled, cross-over design.

Hypothesis 1: Intranasal insulin improves acutely regional perfusion and vasoreactivity in older patients with T2DM as compared with placebo and compared with the control group.

Hypothesis 2: Intranasal insulin improves cognitive functioning including attention, memory and executive function in diabetic patients as compared with placebo and compared with control group.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a major risk factor for vascular dementia. DM alters insulin transport across blood-brain barrier affecting perfusion and neuronal function. Intranasal administration enables effective delivery of insulin to the brain. Clinical studies demonstrated improvement of cognitive function and memory in healthy and cognitively impaired people.

Aim 1: To determine the acute effects of a single 40-IU dose of intranasal insulin vs. placebo on regional perfusion and vasoreactivity to CO2 challenge measured by 3-D continuous arterial spin labeling (CASL) MRI at 3 Tesla in the control and diabetic groups. We will use transcranial Doppler to determine the effects on intranasal insulin vs. placebo on cerebral autoregulation based on measurements of beat-to-beat pressure flow velocity relationship.

Aim 2: To determine whether intranasal insulin improves cognitive functioning in older T2DM patients as compared with placebo and the control group.

This translational study will address an important area about the effects of intranasal insulin on cerebral blood flow regulation and cognition in older diabetics that has not been studied. Intranasal insulin administration may provide a novel therapeutic target for prevention and treatment of microvascular disease and cerebrovascular complications of T2DM. If successful, this approach may have significant impact on the clinical management of large population of older adults with T2DM.

ELIGIBILITY:
Inclusion Criteria:

Diabetes group:

* 30 men and women aged >50 years old diagnosed with T2DM and treated > 5 years with oral agents
* Diabetes severity will be assessed from diabetes duration, hemoglobin A1C, and fasting glucose levels.

Control group:

* 30 healthy men and women aged >50 years selected to have the same age and sex distributions as the diabetic subjects
* Normotensive, not treated for any systemic disease, and have normal fasting blood glucose.

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* History of severe hypoglycemia or hypoglycemic episode during home baseline monitoring
* Positive stress test for CAD or other ischemic conditions
* Carotid stenosis > 50% by medical history
* History of a clinically documented stroke
* Treatment with any medications administered intranasally including intranasal steroids
* Any previous adverse or allergic reactions to insulin
* Acute or unstable medical condition including Myocardial infarction or major illness and surgery within six months
* Liver or renal failure or transplant
* Uncontrolled hypertension (systolic BP >180 and/or diastolic BP >100 mm Hg or subjects taking more than 3 antihypertensive medications)
* Seizure disorders
* Malignant tumors
* Clinical dementia (by history) or inability to follow details of the protocol(MMSE (Mini Mental Status Exam) score (≥3 points below the Comparative Normal Value for the subject's age group and education level, or ≤ 24)
* Current recreational drug or alcohol abuse
* Morbid obesity (BMI >40)
* Inability to obtain permission for participation from the primary care physician
* Transcranial Doppler (TCD) exclusion criterion - poor insonation window and TCD signal
* MR exclusion criteria - any metal or bioimplants not compatible with 3 Tesla MRI and claustrophobia
* Clinically significant and movement limiting hip, knee and/or back disorders or injury, and rheumatoid arthritis

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Novak, MD PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Novak V, Milberg W, Hao Y, Munshi M, Novak P, Galica A, Manor B, Roberson P, Craft S, Abduljalil A. Enhancement of vasoreactivity and cognition by intranasal insulin in type 2 diabetes. Diabetes Care. 2014;37(3):751-9. doi: 10.2337/dc13-1672. Epub 2013 Oct 7. PMID 24101698
- [Result] Zhang H, Hao Y, Manor B, Novak P, Milberg W, Zhang J, Fang J, Novak V. Intranasal insulin enhanced resting-state functional connectivity of hippocampal regions in type 2 diabetes. Diabetes. 2015 Mar;64(3):1025-34. doi: 10.2337/db14-1000. Epub 2014 Sep 23. PMID 25249577

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty consented subjects, 15 type 2 diabetic and 14 controls completed the protocol. One control was excluded after starting the study. Screened participants that did not start study: 27 were excluded after screening visit, 7 withdrew consent. Enrollment Table list the characteristics of 29 participants who completed the protocol.
Groups:
- Diabetes Group: Placebo First; Diabetes Group: Insulin First; Control Group: Placebo First; Control Group: Insulin First: Comparisons of acute effects of intranasal insulin or placebo on cerebral blood flow and cognition.
  Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo
Period: Overall Study
Arm/Group | Diabetes Group: Placebo First | Diabetes Group: Insulin First | Control Group: Placebo First | Control Group: Insulin First
Started | 4 | 11 | 9 | 6
Completed | 4 | 11 | 9 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Twenty nine consented subjects, 15 type 2 diabetic and 14 controls completed the protocol.
Groups:
- Healthy; Diabetics: Comparisons of acute effects of intranasal insulin or placebo on cerebral blood flow and cognition.
  Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo ( sterilesaline) in type 2 diabetes and the non-diabetic control group.Each participant received a single dose of insulin and a single dose of placebo on 2 consequent days in random order.
- Total: Total of all reporting groups
Arm/Group | Healthy | Diabetics | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.9) | 62.0 (7.9) | 61.1 (8.81)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Outcome: Brief Visuospatial Spatial Memory Test -Total Recall (Unit T Score)
Description: To determine the acute effects of a single 40-IU dose of intranasal insulin vs. placebo on cognition and regional perfusion and vasoreactivity to CO2 challenge measured by 3-D continuous arterial spin labeling (CASL) MRI at 3 Tesla in the control and diabetic groups.
  Cognitive outcome: Brief Visuospatial Spatial Memory test -Total Recall (unit T Score).
  Perfusion outcome: Regional vasoreactivity (ml/100g/min/mmHg).
  Each participant received a single dose of intranasal insulin (INI) or placebo on day 2 and a single dose dose of insulin or placebo on day 3 in a random order.
  Acute effects on baseline perfusion, regional vasoreactivity and cognition were determined within 2 hours after administration of insulin or placebo.
Time Frame: Acute changes within 2 hours
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Diabetes Group: Placebo: Comparisons of acute effects of intranasal insulin or placebo on cerebral blood flow and cognition.
  Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo in type 2 diabetes and the control group on cognitive function (Brief Visuospatial Memory test-Revised (BVMT-R)).
- Diabetes Group: Insulin: Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo in type 2 diabetes and the control group.
- Control Group: Placebo; Control Group: Insulin: Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo in type 2 diabetes and the control group on cognitive function (Brief Visuospatial Memory test-Revised (BVMT-R)).
Arm/Group | Diabetes Group: Placebo | Diabetes Group: Insulin | Control Group: Placebo | Control Group: Insulin
Number analyzed (Participants) | 15 | 15 | 14 | 14
T-score | 39.46 (8.86) | 41.23 (9.85) | 43.1 (17.29) | 50.9 (9.66)

2. Primary Outcome: Perfusion Outcome: Right Insular Cortex Perfusion (ml/100g/Min/mmHg)
Description: To determine the acute effects of a single 40-IU dose of intranasal insulin vs. placebo on cognition and regional perfusion and vasoreactivity to CO2 challenge measured by 3-D continuous arterial spin labeling (CASL) MRI at 3 Tesla in the control and diabetic groups.
  Cognitive outcome: Brief Visuospatial Spatial Memory test -Total Recall (unit T Score).
  Perfusion outcome: Regional vasoreactivity (ml/100g/min/mmHg).
Time Frame: Acute changes within 2 hours
Measure: Mean (Standard Deviation); unit: ml/100g/min/mmHg
Arm/Group | Diabetes Group: Placebo | Diabetes Group: Insulin | Control Group: Placebo | Control Group: Insulin
Number analyzed (Participants) | 15 | 15 | 14 | 14
ml/100g/min/mmHg | 39.2 (3.3) | 46.4 (3.6) | 40.3 (2.4) | 36.9 (2.5)

ADVERSE EVENTS:
Groups:
- Diabetes Group: Placebo; Diabetes Group: Insulin; Control Group: Placebo; Control Group: Insulin: Comparisons of acute effects of intranasal insulin or placebo on cerebral blood flow and cognition.
  Intranasal insulin: The acute effects of a single 40-IU dose of intranasal insulin vs. placebo in type 2 diabetes and the non-diabetic control group.
  The intranasal administration of insulin was safe, with no serious adverse events or hypoglycemic episodes and the protocol was feasible for participants.
Arm/Group | Diabetes Group: Placebo | Diabetes Group: Insulin | Control Group: Placebo | Control Group: Insulin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Group: Placebo (N=15) | Diabetes Group: Insulin (N=15) | Control Group: Placebo (N=15) | Control Group: Insulin (N=15)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Healthy-Insulin : One control subject was identified to have un-diagnosed hypertension prior and after intranasal insulin administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No